CLINICAL TRIAL: NCT02308865
Title: Impact of Early Palliative Care on Quality of Life and Survival of Patients With Non-small-cell Metastatic Lung Cancer in Northern France
Brief Title: Early Palliative Care in Metastatic Lung Cancer in Northern France
Acronym: IMPAQ
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor decision
Sponsor: University Hospital, Lille (Other)
Collaborators: Santelys Association (Other); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013_70; 2014-A00514-43 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Lung Cancer Metastatic
Keywords: Early palliative care; Lung cancer; Quality of life
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Patient supported by the onco respiratory service for the treatment of their disease by chemotherapy and for the treatment of complications.
- intervention arm (Experimental): Multi disciplinary palliative care monthly consultations with a doctor, a nurse, a psychologist and posibility of a physical therapist and a chaplain in addition to standard onco-pneumologic care.
  Interventions: Other: multi disciplinary palliative care monthly consultations

INTERVENTIONS:
Other: multi disciplinary palliative care monthly consultations — multi disciplinary palliative care consultations with a doctor, a nurse, a psychologist and posibility of a physical therapist and a worship person.The primary consultation within 3 weeks inclusion and then every month at the same time that consultations onco-respiratory
  Arms: intervention arm

SUMMARY:
Single-center, prospective, controlled, open-label, randomized, two parallel arms comparing early Palliative care versus Standard care in patients with non-small-cell metastatic lung cancer

DETAILED DESCRIPTION:
144 patients will be included; 72 per arm.

* "Standard" Control arm: patient supported by the onco-respiratory service.
* Intervention arm: patients benefit from early palliative care in addition to standard onco-pneumologic care.

The main criterion of judgment is the TOI score measured at 12 weeks.

FACTL questionnaires, HADS and PHQ-9 will be filled out before randomization , at 12 weeks and 21 weeks

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with non-small cell lung cancer

  * Proven histologically
  * Metastatic proven imaging (MRI, CT Scanner, PET scan)
  * Stage IV (any T, any N, M1)
* prior to secondary chemotherapy treatment.
* Age> 18 years
* PS ≤2
* Patient able to understand the nature, purpose and methodology of the study
* signed Informed consent

Exclusion Criteria:

* Age <18 years
* Patient already supported by palliative care
* Patient with an activating EGFR mutation or EML4-ALK rearrangement or ROS1 gene translocation
* Patient under trusteeship / guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-10-17 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
quality of life | 12 weeks
  quality of life is measured at 12 weeks by the TOI score

SECONDARY OUTCOMES:
SURVIVAL | from baseline
EVENTS | 14 days before deaths
  presence of any of the following: chemotherapy, use of resuscitation or no treatment limiting decision 14 days before deaths
QUALITY OF LIFE | 12 and 21 weeks
  quality of life is measured by the score TOI at 12 weeks and by the Echelle SCNS - SF34 scale, FACTL, PHQ-9 and HADS questionnaires at 12 and 21 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Licia Touzet, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU, Hôpital Claude Huriez, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875